CLINICAL TRIAL: NCT06334159
Title: Guided Bone Regeneration Using Fixed vs Non-Fixed Resorbable Collagen Membranes: A Randomized Controlled Clinical Trial
Brief Title: Guided Bone Regeneration Using Fixed vs Non-Fixed Resorbable Collagen Membranes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2019-08
Record Dates: First submitted 2024-02-19; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: non fixed resorbable collagen membranes (control group), versus fixed resorbable collagen membranes (test group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Horizontal Guided Bone Regeneration with a mixture of xenograft (Cerabone 0.5-1mm particles) and allograft (Maxgarft <2mm particles) bone substitute (50/50) with non-fixed resorbable collagen membranes (Jason Membrane 20x30mm)
  Interventions: Procedure: Horizontal GBR without the use of non-resorbable pins for the stabilization of the collagen membrane
- Test Group (Experimental): Horizontal Guided Bone Regeneration with a mixture of xenograft (Cerabone 0.5-1mm particles) and allograft (Maxgarft <2mm particles) bone substitute (50/50) with fixed resorbable collagen membranes(Jason Membrane 20x30mm) with the use of pins (Titan Pins)
  Interventions: Procedure: Horizontal GBR with the use of non-resorbable pins for the stabilization of the collagen membrane

INTERVENTIONS:
Procedure: Horizontal GBR with the use of non-resorbable pins for the stabilization of the collagen membrane — Horizontal Guided Bone Regeneration, with a mixture of xenograft (Cerabone®) and allograft (Maxgraft®), on a 50-50 mixture ratio, grafted in the area required to be augmented, and then covered by a collagen membrane (Jason® membrane), being fixed with non-resorbable pins (Test Group).
  Arms: Test Group
Procedure: Horizontal GBR without the use of non-resorbable pins for the stabilization of the collagen membrane — Horizontal Guided Bone Regeneration, with a mixture of xenograft (Cerabone®) and allograft (Maxgraft®), on a 50-50 mixture ratio, grafted in the area required to be augmented, and then covered by a collagen membrane (Jason® membrane), being left unfixed (Control Group).
  Arms: Control Group

SUMMARY:
The aim of this clinical trial is to compare the horizontal bone gain when grafting a bone substitute with non fixed resorbable collagen membranes (control group), versus fixed resorbable collagen membranes (test group) in resorbed ridges requiring Guided Bone Regeneration (GBR) to facilitate implant placement at 6 months.

DETAILED DESCRIPTION:
The aim of this clinical trial is to compare the horizontal bone gain when grafting a mixture of xenograft and allograft (50/50) with non fixed resorbable collagen membranes (control group), versus fixed resorbable collagen membranes (test group) in resorbed ridges requiring Guided Bone Regeneration (GBR) to facilitate implant placement at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years old or older
2. Patients requiring Guided Bone Regeneration due to insufficient ridge width(≤5mm) to place dental implants, with sufficient vertical ridge height (≥9mm) from vital anatomical structures (the inferior alveolar nerve in the Mandible, or the sinus in the Maxilla)
3. One or more teeth missing in posterior zone (Premolars, and Molars)
4. Absence of active Periodontal disease
5. Good level of oral hygiene (Plaque index <25%)
6. Absence of systemic diseases that could influence the outcome of the therapy (Uncontrolled diabetes, osteoporosis, bisphosphonate medications)
7. Non smokers or light smokers (<10 cigarettes per day)
8. Informed consent signed

Exclusion Criteria:

1. Patients with sufficient ridge width (>5 mm) and height (≥9mm) from vital anatomical structure) requiring no GBR to place dental implants
2. Patients with severe horizontal and vertical defects requiring other surgical techniques.
3. Long-term non-steroidal anti-inflammatory drug therapy (3months).
4. Lactating females or currently pregnant women.
5. Severe cognitive or psychiatric disorders.
6. Unwillingness to return for follow-up examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Horizontal Bone Gain | T3: 6 months after the Horizontal GBR
  To compare the horizontal bone gain when grafting a mixture of xenograft and allograft (50/50) with non-fixed resorbable collagen membranes (control group) versus fixed resorbable collagen membranes (test group) in resorbed ridges requiring GBR to facilitate implant placement at 6 months.
  Along the 6 months, 3 Cone Beam Computed Tomography scans (CBCT) will be needed. At baseline (T1), the first CBCT will be taken before performing any surgical procedure to measure the initial width of the ridge. Immediately after the GBR (T2), a second CBCT scan will be taken, which will be useful to measure new ridge width in each group. Finally, at 6 month follow-up a third CBCT scan will be taken (T3) in order to assess the difference with T1 regarding amount of bone gain horizontally, and with T2 regarding horizontal dimensional stability of the grafted bone in each of the 2 groups.
Bone Width Gain | T3: 6 months after the Horizontal GBR
  To compare the bone width gain between the test group and control group, 6 months after the horizontal GBR.
  A caliper will be used in order to evaluate and compare the bone width gain at T1, T2, and T3 between the Test and Control Groups. These measurements are performed intra-operatively before the Horizontal GBR (T1), immediately after (T2), and at 6 months (T3) at the time of implant placement. Measurements will be performed at 1cm, 3cm, and 5cm apical from the bone crest at the regenerated area.

SECONDARY OUTCOMES:
Horizontal Dimensional Stability | T3: 6 months after the Horizontal GBR
  To compare the horizontal dimensional stability of the augmented ridges between the test group and control group after 6 months.
  After the surgical procedure, a CBCT scan (T2) will be completed and the bone width will be assessed and compared with the bone width at 6 months postoperatively when a new CBCT scan (T3) will be completed before implant placement.
Post-surgical complications | T2-T3: From the surgery to 6 months
  To compare the post-surgical complications that may occur between the test group and control group throughout the period of healing and during the following 6 months. The complications will be evaluated using the Healing Complications Classification, as suggested by Fontana et al. 2011. The healing post-surgical complications are divided into four classes, according to the presence and extent of exposure, as well as the presence of a purulent exudate:
  * Class I: membrane exposure <3mm, no purulent exudate
  * Class II: membrane exposure ≥3mm, no purulent exudate
  * Class III: membrane exposure with purulent exudate
  * Class IV: abscess, without membrane exposure
Patient's satisfaction | At 2-weeks follow up after the surgical procedure
  To compare patient's satisfaction regarding the post-operative pain and compare it between the test group and control group throughout the period of healing and during the following 6 months, through the use of a Visual Analogue Scale (VAS). It is a 10cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patients will be asked to mark their average experience of discomfort and pain. The scores of the VAS will be obtained by measuring the distance in centimeters (0 to 10).
Histologic examination of the augmented bone at 6 months | At time of implant placement
  To examine type of cells present after 6 months of procedure by performing histological examination to the sample harvested from the site with the use of an implant trephine drill. The histologic evaluation will be performed in order to evaluate the type of cells present at the site of augmentation

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Vallés, DDS, MS, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Georgios Markantonatos, Barcelona, Sant Cugat Del Vallès, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pagni G, Pellegrini G, Giannobile WV, Rasperini G. Postextraction alveolar ridge preservation: biological basis and treatments. Int J Dent. 2012;2012:151030. doi: 10.1155/2012/151030. Epub 2012 Jun 12. PMID 22737169
- [Background] Paolantonio M, Dolci M, Scarano A, d'Archivio D, di Placido G, Tumini V, Piattelli A. Immediate implantation in fresh extraction sockets. A controlled clinical and histological study in man. J Periodontol. 2001 Nov;72(11):1560-71. doi: 10.1902/jop.2001.72.11.1560. PMID 11759868
- [Background] Hua Wang, Chunfu Deng, Baohong Zhao, Dehao Shang, Chong Zhang, The Effect of Bone Formation with Bio-Oss Guided by Collagen Membrane, Journal of Hard Tissue Biology, 2013, 22 巻, 2 号, p. 255-260, 公開日 2013/04/26, Online ISSN 1880-828X, Print ISSN 1341-7649, https://doi.org/10.2485/jhtb.22.255, https://www.jstage.jst.go.jp/article/jhtb/22/2/22_255/_article/-char/ja, 抄録
- [Background] Lee SW, Kim SG. Membranes for the Guided Bone Regeneration. Maxillofac Plast Reconstr Surg. 2014 Nov;36(6):239-46. doi: 10.14402/jkamprs.2014.36.6.239. Epub 2014 Nov 12. PMID 27489841
- [Background] Dimitriou R, Mataliotakis GI, Calori GM, Giannoudis PV. The role of barrier membranes for guided bone regeneration and restoration of large bone defects: current experimental and clinical evidence. BMC Med. 2012 Jul 26;10:81. doi: 10.1186/1741-7015-10-81. PMID 22834465
- [Background] Urban IA, Lozada JL, Wessing B, Suarez-Lopez del Amo F, Wang HL. Vertical Bone Grafting and Periosteal Vertical Mattress Suture for the Fixation of Resorbable Membranes and Stabilization of Particulate Grafts in Horizontal Guided Bone Regeneration to Achieve More Predictable Results: A Technical Report. Int J Periodontics Restorative Dent. 2016 Mar-Apr;36(2):153-9. doi: 10.11607/prd.2627. PMID 26901293
- [Background] Amano Y, Ota M, Sekiguchi K, Shibukawa Y, Yamada S. Evaluation of a poly-l-lactic acid membrane and membrane fixing pin for guided tissue regeneration on bone defects in dogs. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Feb;97(2):155-63. doi: 10.1016/j.tripleo.2003.09.009. PMID 14970774
- [Background] Francis J. Hughes. Stem Cell Biology and Tissue Engineering in Dental Sciences, Academic Press,2015, ISBN 9780123971579: 434-444
- [Result] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Result] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Result] Cucchi A, Vignudelli E, Napolitano A, Marchetti C, Corinaldesi G. Evaluation of complication rates and vertical bone gain after guided bone regeneration with non-resorbable membranes versus titanium meshes and resorbable membranes. A randomized clinical trial. Clin Implant Dent Relat Res. 2017 Oct;19(5):821-832. doi: 10.1111/cid.12520. Epub 2017 Jul 26. PMID 28745035
- [Result] Sisti A, Canullo L, Mottola MP, Covani U, Barone A, Botticelli D. Clinical evaluation of a ridge augmentation procedure for the severely resorbed alveolar socket: multicenter randomized controlled trial, preliminary results. Clin Oral Implants Res. 2012 May;23(5):526-35. doi: 10.1111/j.1600-0501.2011.02386.x. Epub 2011 Dec 8. PMID 22150876